CLINICAL TRIAL: NCT00801073
Title: Comparison Amongst Scleral, Corneal and Amniotic Membrane Grafts to Restore Scleral Thinning
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Jose Alvaro Pereira Gomes, Departamento de Oftalmologia/Instituto da Visão, Universidade Federal de São Paulo (UNIFESP), Brazil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0060 / 04
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2008-12-03 (Estimated); Status verified 2008-12

CONDITIONS: Scleral Thinning
Keywords: Amniotic membrane; Cornea; Scleral thinning
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amniotic Membrane Transplantation (Experimental): Human Amniotic Membrane Transplantation for The Treatment of Ocular Surface Disease
  Interventions: Procedure: Human Amniotic Membrane Transplantation

INTERVENTIONS:
Procedure: Human Amniotic Membrane Transplantation — Human Amniotic Membrane Transplantation for The Treatment of Ocular Surface Disease

SUMMARY:
The purpose of this study is to evaluate the use of preserved scleral, corneal and amniotic membrane graft for the surgical repair of scleral thinning of different sizes in patients underwent surgery of pterygium with associated beta therapy .

DETAILED DESCRIPTION:
Scleral thinning may occur secondary to different ocular surface conditions, especially in rheumatologic diseases and after surgeries as in pterygium. There are different methods to treat this condition, as to use scleral, corneal and more recently amniotic membrane graft.

ELIGIBILITY:
Inclusion Criteria:

* Patients with corneal scleral defects that have persisted for 1 years or longer, regardless of their cause. These patients will have received corneal-scleral or amniotic membrane transplant in order to correct scleral thinning
* Patients with history of pterygium surgery associated with beta therapy followed by scleral thinning

Exclusion Criteria:

* Ocular infection
* Acute ocular inflammatory condition
* Previous ocular surgery in the eye study
* Non-controlled systemic disease such as rheumatoid arthritis

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-02; Primary Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
The surgical procedure was randomized in scleral, corneal or amniotic membrane graft. Nine patients underwent surgery with scleral graft that was covered by conjunctival flap; ten with corneal graft and ten with amniotic membrane transplantation. | Patients were followed for 180 days.